CLINICAL TRIAL: NCT01111968
Title: Evaluation of Safety, Tolerability and Immunogenicity of Adjuvanted Candidate Vaccines Against Pandemic Influenza A (H1N1)
Brief Title: Evaluation of Pandemic Influenza A (H1N1)Candidate Vaccines
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Butantan Institute (Other Government)
Collaborators: Hospital Universitario da USP (Unknown); University of Sao Paulo (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: BUTVAC - Influenza A (H1N1)
Record Dates: First submitted 2010-04-14; First posted 2010-04-28 (Estimated); Last update posted 2013-02-06 (Estimated); Status verified 2013-02

CONDITIONS: Influenza
Keywords: vaccine; pandemic influenza A; adjuvant; safety
MeSH Terms: conditions — Influenza, Human | interventions — hexavalent group A streptococcal vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (10):
- pandemic vaccine 1 (Experimental): 7,5µg of A/H1N1 with MPLA adjuvant - IB, suspension (5µg) + Al(OH)3
  Interventions: Biological: pandemic vaccine 1
- pandemic vaccine 2 (Experimental): 3,75µg of A/H1N1 with MPLA adjuvant - IB, suspension (5µg) + Al(OH)3
  Interventions: Biological: pandemic vaccine 2
- pandemic vaccine 5 (Experimental): 7,5µg of A/H1N1 with MPLA adjuvant - IB, emultion (5µg) + Al(OH)3 + Squalene 2% emulsion
  Interventions: Biological: pandemic vaccine 5
- pandemic vaccine 6 (Experimental): 3,75µg of A/H1N1 with MPLA adjuvant - IB, emultion (5µg) + Al(OH)3 + Squalene 2% emultion
  Interventions: Biological: pandemic vaccine 6
- pandemic vaccine 9 (Experimental): 7,5 µg of A/H1N1 with Al(OH)3 + Squalene 2% emultion
  Interventions: Biological: pandemic vaccine 9
- pandemic vaccine 10 (Experimental): 3,75 µg of A/H1N1 with Al(OH)3 + Squalene 2% emultion
  Interventions: Biological: pandemic vaccine 10
- pandemic vaccine 11 (Experimental): 7,5µg of A/H1N1 with Al(OH)3
  Interventions: Biological: pandmeic vaccine 11
- pandemic vaccine 12 (Experimental): 3,75µg of A/H1N1 with Al(OH)3
  Interventions: Biological: pandmeic vaccine 12
- pandemic vaccine 13 (Experimental): 15µg of A/H1N1 with no adjuvant
  Interventions: Biological: pandmic vaccine 13
- placebo group 14 (Placebo Comparator): placebo
  Interventions: Biological: placebo group 14

INTERVENTIONS:
Biological: pandemic vaccine 1 — 7,5µg of A/H1N1 with MPLA adjuvant - IB, suspension (5µg) + Al(OH)3
  Other Names: vaccine group C
  Arms: pandemic vaccine 1
Biological: pandemic vaccine 2 — 3,75µg of A/H1N1 with MPLA adjuvant - IB, suspension (5µg) + Al(OH)3
  Other Names: vaccine group I
  Arms: pandemic vaccine 2
Biological: pandemic vaccine 5 — 7,5µg of A/H1N1 with MPLA adjuvant - IB, emultion (5µg) + Al(OH)3 + Squalene 2% emulsion
  Other Names: vaccine group N
  Arms: pandemic vaccine 5
Biological: pandemic vaccine 6 — 3,75µg of A/H1N1 with MPLA adjuvant - IB, emultion (5µg) + Al(OH)3 + Squalene 2% emultion
  Other Names: vaccine group A
  Arms: pandemic vaccine 6
Biological: pandemic vaccine 9 — 7,5 µg of A/H1N1 with Al(OH)3 + Squalene 2% emultion
  Other Names: vaccine group F
  Arms: pandemic vaccine 9
Biological: pandemic vaccine 10 — 3,75 µg of A/H1N1 with Al(OH)3 + Squalene 2% emultion
  Other Names: vaccine group L
  Arms: pandemic vaccine 10
Biological: pandmeic vaccine 11 — 7,5µg of A/H1N1 with Al(OH)3
  Other Names: vaccine group E
  Arms: pandemic vaccine 11
Biological: pandmeic vaccine 12 — 3,75µg of A/H1N1 with Al(OH)3
  Other Names: vaccine group K
  Arms: pandemic vaccine 12
Biological: pandmic vaccine 13 — 15µg of A/H1N1 with no adjuvant
  Other Names: vaccine group H
  Arms: pandemic vaccine 13
Biological: placebo group 14 — All elements of the vaccine but antigen and adjuvant
  Other Names: vaccine group B
  Arms: placebo group 14

SUMMARY:
This is a prospective phase I study to evaluate the safety, tolerability and immunogenicity of nine adjuvanted candidate vaccines against pandemic influenza A (H1N1) virus.

DETAILED DESCRIPTION:
The candidate vaccines are produced by Butantan institute - Sao Paulo, Brazil

ELIGIBILITY:
Inclusion Criteria:

* Health adults of both genders
* Age ≥ 18 ≤ 50 years
* Able to understand every required study procedure
* Female volunteers should agree to take an acceptable contraceptive method Menopause is characterized by absence of menstrual flux for two consective years
* Normal values for pre-stablished laboratory assays
* Accpetance to participate and sign the consent form

Exclusion Criteria:

* Any chronic condition
* Be on immunossupressive or stimulant therapy
* Have egg alergy
* Have past history of alergy to sazonal influenza vaccine
* Have received another inactivated vaccine within the prior 2 weeks or a live vaccine in the past four weeks to his/her participation in the study
* Acute infectious disease during seven days prior vaccination
* Female on breasthfeeding
* Confirmed prior infection by pandemic influenza A
* Participation in another clinical trial in the last 6 months
* Any other condition identified by the principal investigator which is considered not safe for enrollment of the volunteer

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 266 (Actual)
Dates: Start 2010-01; Primary Completion 2010-12 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
the proportion of subjects with antibody titers of 1:40 or more on hemagglutination-inhibition assay | 21 days after each vaccination
  Volunteers will receive two doses of vaccine,21 days apart.

SECONDARY OUTCOMES:
Safety and tolerability | 30 minutes and 72 hours after vaccination
  Evaluation of local and systemic adverse effects throught the study period

CONTACTS AND LOCATIONS:
Overall Officials: Lucia MA Campos, MD. PhD, Principal Investigator — Children´s Institute - School of Medicine of University of Sao Paulo
Locations (2):
- Brazil (2):
  - Centro de Pesquisa Clinica do Instituto da Criança do hospital das Clinicas da Faculdade de Medicina da USP, São Paulo, São Paulo
  - Centro de Pesquisa Clínica do Hospital Universitário da USP, São Paulo, São Paulo

REFERENCES:
- [Derived] Precioso AR, Miraglia JL, Campos LM, Goulart AC, Timenetsky Mdo C, Cardoso MR, Luna E, Mondini G, Guedes Jda S, Raw I. A phase I randomized, double-blind, controlled trial of 2009 influenza A (H1N1) inactivated monovalent vaccines with different adjuvant systems. Vaccine. 2011 Nov 8;29(48):8974-81. doi: 10.1016/j.vaccine.2011.09.040. Epub 2011 Sep 21. PMID 21945258